CLINICAL TRIAL: NCT04208204
Title: Somatocognitive Therapy in Treatment of Provoked Vestibulodynia - Process of Change and User Experience
Brief Title: Somatocognitive Therapy in Treatment of Provoked Vestibulodynia - a Feasibility Study
Acronym: ProLoVe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo Metropolitan University (Other)
Collaborators: Oslo University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2018/1036
Record Dates: First submitted 2019-10-30; First posted 2019-12-23 (Actual); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: Provoked Vestibulodynia
Keywords: provoked localized vulvodynia; provoked vestibulodynia; vestibulitt; physiotherapy

STUDY DESIGN:
Intervention Model Description: Three measurements time points: baseline, after treatment, and 8 months after baseline. Additionally two interviews per participant; first - between baseline and treatment ending and second after 8 months follow up
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Somatocognitive physiotherapy (Experimental): Every participant will maximally receive 15 individual sessions of somatocognitive physiotherapy
  Interventions: Other: somatocognitive physiotherapy

INTERVENTIONS:
Other: somatocognitive physiotherapy — Somatocognitive physiotherapy (SCT) is a multimodal physical therapy approach that has been developed in an attempt at alleviating the burden of longstanding pain. The main foci of SCT include: (1) bodily exercises and techniques increasing body awareness, ability to relax and control muscle tension in different situations; (2) education about the vulvodynia and factors influencing pain experience; (3) coping with emotions and thoughts related to bodily experiences; and (4) structured homework assignments promoting application of the learned techniques in daily situation and gradual exposure to activities associated with pain. An important goal of SCT is to facilitate integration of new bodily habits into the patient's daily activities. The most important learning process thus occurs in the space between the treatment sessions. The therapeutic techniques are to be rehearsed in everyday situations.

SUMMARY:
This study examines feasibility of R&D activities in the planned randomized controlled trial where effectiveness of somatocognitive therapy intervention will be compared to treatment as usual in provoked vestibulodynia.

DETAILED DESCRIPTION:
Provoked vestibulodynia is a multifactorial, persistent pain condition, affecting young women. It represents the most common cause of pain during sexual intercourse. Existing treatment approaches are predominantly based on clinical experience, observational studies, or reports of expert committees. Although, physiotherapy is one of the most commonly recommended treatments, high quality randomized controlled trials are needed to assess its effectiveness.

This is a phase I, feasibility study with the purpose of testing R&D activities for a planned full size RCT. Additionally, patients experiences with the somatocognitive therapy intervention, assessment measures and condition itself will be collected using qualitative interviews. The results will be applied to adjust time-line of the treatment, outcome measures and therapeutic approach before commencing full scale RCT.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed provoked vestibulodynia diagnosis

Exclusion Criteria:

* vulvar pain is not clearly linked to intercourse or pressure applied to vestibule or usage of tampon
* active infection or dermatologic lesion in the vulvar region

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | 5 months
  Number of eligible patients and number of recruited participants per week
Follow-up rate | 8 months
  The follow-up rate is measured by the percentage of participants who were followed up successfully until the 8 months follow-up
Adherence | 8 months
  Adherence is defined as the number of participants who fully complete the battery of self-report questionnaires, 14-day diary, biweekly forms about the received treatment and perform Tampon tests.
Evaluation of Tampon test as a primary outcome measure - score variance | 8 months
  Participants perform Tampon test 3 times in course of 14 days (day1, 7 and 14) at each of the 3 time points (baseline, post-treatment, 8 months after baseline), 9 scores in total. Numerical rating scale (0-10) will be used to score pain intensity. Intra-individual score variance will be estimated as difference between the min and max score at each time point for every participant. Lower variability is better.
Adverse events | 8 months
  If participant is pulled out of the study because somatocognitive therapy is deemed as a non-appropriate treatment (e.g. participant is instead referred to psychological counselling), such event is recorded as adverse.
Evaluation of Tampon test as a primary outcome measure - qualitative interviews | 8 months
  All participants are asked in individual qualitative interviews if they experience a Tampon test as a relevant instrument for assessing pain sensitivity experienced during intercourse.

SECONDARY OUTCOMES:
Implementation and acceptability of the somatocogntive therapy intervention | 8 months
  Participants will be asked in qualitative interviews about their experiences with somatocogntitve therapy intervention. Global Rating of Change scale will be used to provide quantitative estimation of participants' satisfaction with the treatment effect directly after treatment and at 8 months follow-up. The scale ranges from 1 to 6. Score of 1 means that treatment helped a lot and the score of 6 means that the treatment made the condition much worse.
Evaluation of somatocognitive therapy intervention's potential to reduce pain | 8 months
  Changes in individual mean scores (0-10, the lower score the better) of pain experienced during tampon test between 3 measurements time points.
Evaluation of somatocognitive therapy intervention's potential to improve sexual functioning | 8 months
  Changes in individual scores on Female Sexual Function Index between 3 measurements time points. Scale ranges 0-36, higher score means better sexual functioning.
Evaluation of somatocognitive therapy intervention's potential to reduce psychological distress | 8 months
  Changes in individual scores on Hopkins Symptom Check List - 25 questions version between 3 measurements time points. Scale ranges 1-4, lower score indicates less psychological distress.
Evaluation of somatocognitive therapy intervention's potential to reduce pain catastrophizing | 8 months
  Changes in individual scores on Pain Catastrophizing Scale between 3 different time points. Scale ranges 0-52, the lower score represents less pain catastrophizing

CONTACTS AND LOCATIONS:
Overall Officials: Slawomir Wojniusz, PhD, Principal Investigator — Oslo Metropolitan University
Locations (1):
- Oslo Metropolitan University, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kaarbo MB, Danielsen KG, Haugstad GK, Helgesen ALO, Wojniusz S. Feasibility and acceptability of somatocognitive therapy in the management of women with provoked localized vestibulodynia-ProLoVe feasibility study. Pilot Feasibility Stud. 2022 Mar 23;8(1):68. doi: 10.1186/s40814-022-01022-2. PMID 35321744
- [Derived] Kaarbo MB, Danielsen KG, Haugstad GK, Helgesen ALO, Wojniusz S. The Tampon Test as a Primary Outcome Measure in Provoked Vestibulodynia: A Mixed Methods Study. J Sex Med. 2021 Jun;18(6):1083-1091. doi: 10.1016/j.jsxm.2021.03.010. Epub 2021 May 6. PMID 33967000